CLINICAL TRIAL: NCT01758861
Title: Effect of Erythropoietin on the Incidence of Acute Kidney Injury Following Complex Valvular Heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2011-0355
Record Dates: First submitted 2012-12-17; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Acute Kidney Injury
Keywords: Erythropoietin; acute kidney injury; valvular heart surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPO group (Experimental): EPO group received 300 IU/kg of rHuEPO-alpha via intravenous bolus administration after induction of anesthesia.
  Interventions: Drug: EPO group
- Placebo group (Placebo Comparator): Placebo group received normal saline via intravenous bolus administration after induction of anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EPO group
  Other Names: EPO group received 300 IU/kg of rHuEPO-alpha via intravenous bolus administration after induction of anesthesia.
  Arms: EPO group
Drug: Placebo
  Arms: Placebo group

SUMMARY:
Acute kidney injury (AKI) frequently occurs after cardiac surgery using cardiopulmonary bypass (CPB). Recombinant human erythropoietin (rHuEPO) is known to provide organ protection against ischemia-reperfusion injury through its anti-inflammatory properties. The aim of the present study was to investigate the effect of a single preoperative bolus of EPO on the incidence of AKI following complex valvular heart surgery in a randomized, controlled and double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

* preoperative risk factors for AKI and scheduled for complex valvular heart operations
* Enrolled criteria for high risk of AKI were patients with more than 2 of bellows: female, serum creatinine >1.2 mg/dl, preoperative A-fib, GFR < 60 ml/min, NYHA class IV, HTN, DM, age > 65 years, peripheral vascular disease.
* Complex valvular heart operations were defined as double-valve surgery, combined valve and coronary artery bypass grafting procedures, Bentall operation, combined mitral valve surgery and tricuspid annuloplasty or reoperation.

Exclusion Criteria:

* Patients with preexisting uncontrolled hypertension (diastolic blood pressure > 100 mmHg), immunosuppression, history of thromboembolism, malignant disease, seizure, liver dysfunction, renal impairment (serum creatinine > 2 mg/dL), and drug or alcohol abuse were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
incidence of acute kidney injury | change of renal function including SCr, cystatin C, creatinine clearance from 24 h before operation to postoperative day (POD) 5
  The diagnostic criteria for AKI is followed by AKIN criteria (absolutely increase in the SCr concentration ≥ 0.3 mg/dL from baseline, ≥ 50% increase in the SCr concentration within 48 hours after operation).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesiology and pain medicine Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JH, Shim JK, Song JW, Song Y, Kim HB, Kwak YL. Effect of erythropoietin on the incidence of acute kidney injury following complex valvular heart surgery: a double blind, randomized clinical trial of efficacy and safety. Crit Care. 2013 Oct 24;17(5):R254. doi: 10.1186/cc13081. PMID 24156702